CLINICAL TRIAL: NCT03669302
Title: Activity-Dependent Transspinal Stimulation for Recovery of Walking Ability After Spinal Cord Injury
Brief Title: Activity-Dependent Transspinal Stimulation in SCI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID
Sponsor: City University of New York (Other)
Collaborators: Bronx Veterans Medical Research Foundation, Inc (Other)
Responsible Party: Principal Investigator, Maria Knikou, PT, PhD, Professor, City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C33276GG
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Spinal Cord Injuries; Paraplegia, Spinal; Tetraplegia/Tetraparesis; Paraplegia, Spastic
Keywords: locomotor training; transcutaneous spinal cord stimulation; Lokomat; brain stimulation; peripheral nerve stimulation; H-reflex; spinal neural circuits; neuroplasticity; recovery
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Quadriplegia

STUDY DESIGN:
Intervention Model Description: Individuals with Spinal Cord Imjury will be randomly assigned to receive robotic gait training with the Lokomat, and/or Lokomat gait training combined with non-invasive thoracolumbar transspinal stimulation at 0.3 or at 30 Hz.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Robotic gait training (Sham Comparator): Robotic gait training only
  Interventions: Other: Robotic gait training
- Robotic gait training & low-frequeny transspinal stimulation. (Experimental): Robotic gait training will be administered along with non-invasive transspinal stimulation over the thoracolumbar region during assisted stepping at low frequency (0.3 Hz).
  Interventions: Device: Robotic gait training and low-frequency transspinal stimulation
- Robotic gait training & high-frequeny transspinal stimulation. (Experimental): Robotic gait training will be administered along with non-invasive transspinal stimulation over the thoracolumbar region during assisted stepping at high frequency (30 Hz).
  Interventions: Device: Robotic gait training and high-frequency transspinal stimulation

INTERVENTIONS:
Other: Robotic gait training — Fifteen people with spinal cord injury will receive 20 daily sessions of robotic gait training. During assisted stepping, they will receive also non-invasive transspinal stimulation as a pulse train at 30 Hz during the stance phase of gait. Before and after training standardized clinical and neurophysiological tests will be used to assess recovery of sensorimotor function.
  Arms: Robotic gait training
Device: Robotic gait training and low-frequency transspinal stimulation — Fifteen people with spinal cord injury will receive 20 daily sessions of robotic gait training. During assisted stepping, they will receive also non-invasive transspinal stimulation as a single pulse at 0.3 Hz during the stance phase of gait. Before and after training standardized clinical and neurophysiological tests will be used to assess recovery of sensorimotor function.
  Arms: Robotic gait training & low-frequeny transspinal stimulation.
Device: Robotic gait training and high-frequency transspinal stimulation — Fifteen people with spinal cord injury will receive 20 daily sessions of robotic gait training. During assisted stepping, they will receive also non-invasive transspinal stimulation as a pulse train at 30 Hz during the stance phase of gait. Before and after training standardized clinical and neurophysiological tests will be used to assess recovery of sensorimotor function.
  Arms: Robotic gait training & high-frequeny transspinal stimulation.

SUMMARY:
Robotic gait training is often used with the aim to improve walking ability in individuals with Spinal Cord Injury. However, robotic gait training alone may not be sufficient. This study will compare the effects of robotic gait training alone to robotic gait training combined with either low-frequency or high-frequency non-invasive transspinal electrical stimulation. In people with motor-incomplete SCI, a series of clinical and electrical tests of nerve function will be performed before and after 20 sessions of gait training with or without stimulation.

DETAILED DESCRIPTION:
People with spinal cord injury (SCI) have motor dysfunction that results in substantial social, personal, and economic costs. Robotic gait training is often used with the aim to improve walking ability in these individuals. Investigators recently reported that robotic gait training reorganizes spinal neuronal circuits, improves motor activity, and contributes substantially to recovery of walking ability in people with motor incomplete SCI. However, pathological muscle tone and abnormal muscle activation patterns during assisted stepping were still evident after multiple sessions of robotic gait training. Locomotor training alone may thus be insufficient to strengthen weak neuronal synapses connecting the brain with the spinal cord or to fully optimize spinal neural circuits. On the other hand, spinal cord stimulation increases sprouting and plasticity of axons and dendrites in spinalized animals. Furthermore, transcutaneous spinal cord stimulation (termed here transspinal stimulation) in people with SCI can evoke rhythmic leg muscle activity when gravity is eliminated. A fundamental knowledge gap still exists on induction of functional neuroplasticity and recovery of leg motor function after repetitive thoracolumbar transspinal stimulation during body weight supported (BWS) assisted stepping in people with SCI. The central working hypothesis in this study is that transspinal stimulation delivered during BWS-assisted stepping provides a tonic excitatory input increasing the overall responsiveness of the spinal cord and improving motor output. The investigators will address 3 specific aims: Establish induction of neuroplasticity and improvements in leg sensorimotor function in people with motor incomplete SCI when transspinal stimulation is delivered during BWS-assisted stepping at low frequencies (0.3 Hz; Specific Aim 1) and at high frequencies (30 Hz; Specific Aim 2), and when BWS-assisted step training is administered without transspinal stimulation (Specific Aim 3). In all groups, outcomes after 20 sessions will be measured via state-of-the-art neurophysiological methods. Corticospinal circuit excitability will be measured via transcranial magnetic stimulation motor evoked potentials in seated subjects (Aims 1A, 2A, 3A). Soleus H-reflex and tibialis anterior flexor reflex excitability patterns will be measured during assisted stepping (Aims 1B, 2B, 3B). Sensorimotor function will be evaluated via standardized clinical tests of gait and strength (Aims 1C, 2C, 3C). Additionally, poly-electromyographic analysis of coordinated muscle activation will be measured in detail. It is hypothesized that transspinal stimulation at 30 Hz during assisted stepping improves leg motor function and decreases ankle spasticity more compared to 0.3 Hz. It is further hypothesized that transspinal stimulation at 30 Hz normalizes the abnormal phase-dependent soleus H-reflex and flexor reflex modulation commonly observed during stepping in people with motor incomplete SCI. To test the project hypotheses, 45 people with motor incomplete SCI will be randomly assigned to receive 20 sessions of transspinal stimulation at 0.3 or 30 Hz during BWS-assisted stepping or 20 sessions of BWS-assisted stepping without transspinal stimulation (15 subjects per group). Results from this research project will advance considerably the field of spinal cord research and change the standard of care because there is great potential for development of novel and effective rehabilitation strategies to improve leg motor function after motor incomplete SCI in humans.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of motor incomplete spinal cord injury (SCI).
* SCI is above thoracic 12 vertebra.
* Absent permanent ankle joint contractures.
* SCI occurred 6 months before enrollment to the study.

Exclusion criteria:

* Supraspinal lesions
* Neuropathies of the peripheral nervous system
* Degenerative neurological disorders of the spine or spinal cord
* Motor complete SCI
* Presence of pressure sores
* Urinary tract infection
* Neoplastic or vascular disorders of the spine or spinal cord
* Pregnant women or women who suspect they may be or may become pregnant.
* People with cochlear implants, pacemaker and implanted stimulators
* People with history of seizures
* People with implanted Baclofen pumb

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
Plasticity of cortical and corticospinal neuronal circuits | 3 years
  Neurophysiological tests probing cortical and corticospinal excitability will be measured before and after the intervention. Single-pulse transcranial magnetic stimulation (TMS) will be used to assemble the recruitment curve of motor evoked potentials, and paired-pulse TMS will be used to probe changes in cortical inhibitory and facilitatory neuronal circuits.
Plasticity of spinal neuronal circuits | 3 years
  Neurophysiological tests probing spinal reflex excitability will be measured before and after each intervention by posterior tibial and sural nerves stimulation during Lokomat-assisted stepping depicting the amplitude modulation of the soleus H-reflex and tibialis anterior flexor reflex.

SECONDARY OUTCOMES:
Senorimotor leg motor function | 3 years
  Manual muscle test and leg sensation based on American Spinal Injury Association guidelines.
Spasticity | 3 years
  Tardieu scale
Walking function | 3 years
  Two-minute walk test and 10 meter timed test.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Knikou, PT, PhD, Principal Investigator — Research Foundation of the City University of New York; Noam Y Harel, MD, PhD, Principal Investigator — VA Office of Research and Development
Locations (2):
- United States (2):
  - Department of Physical Therapy, Motor Control and NeuroRecovery Laboratory, Staten Island, New York
  - Veterans Affairs Medical Center, The Bronx, New York

REFERENCES:
- [Background] Marino RJ, Barros T, Biering-Sorensen F, Burns SP, Donovan WH, Graves DE, Haak M, Hudson LM, Priebe MM; ASIA Neurological Standards Committee 2002. International standards for neurological classification of spinal cord injury. J Spinal Cord Med. 2003 Spring;26 Suppl 1:S50-6. doi: 10.1080/10790268.2003.11754575. No abstract available. PMID 16296564
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Adams MM, Ginis KA, Hicks AL. The spinal cord injury spasticity evaluation tool: development and evaluation. Arch Phys Med Rehabil. 2007 Sep;88(9):1185-92. doi: 10.1016/j.apmr.2007.06.012. PMID 17826466
- [Background] Barbeau H, Wainberg M, Finch L. Description and application of a system for locomotor rehabilitation. Med Biol Eng Comput. 1987 May;25(3):341-4. doi: 10.1007/BF02447435. No abstract available. PMID 3449731
- [Background] Carmel JB, Berrol LJ, Brus-Ramer M, Martin JH. Chronic electrical stimulation of the intact corticospinal system after unilateral injury restores skilled locomotor control and promotes spinal axon outgrowth. J Neurosci. 2010 Aug 11;30(32):10918-26. doi: 10.1523/JNEUROSCI.1435-10.2010. PMID 20702720
- [Background] Chang CW, Lien IN. Estimate of motor conduction in human spinal cord: slowed conduction in spinal cord injury. Muscle Nerve. 1991 Oct;14(10):990-6. doi: 10.1002/mus.880141010. PMID 1944412
- [Background] Chen R, Tam A, Butefisch C, Corwell B, Ziemann U, Rothwell JC, Cohen LG. Intracortical inhibition and facilitation in different representations of the human motor cortex. J Neurophysiol. 1998 Dec;80(6):2870-81. doi: 10.1152/jn.1998.80.6.2870. PMID 9862891
- [Background] Colombo G, Wirz M, Dietz V. Driven gait orthosis for improvement of locomotor training in paraplegic patients. Spinal Cord. 2001 May;39(5):252-5. doi: 10.1038/sj.sc.3101154. PMID 11438840
- [Background] Conway BA, Knikou M. The action of plantar pressure on flexion reflex pathways in the isolated human spinal cord. Clin Neurophysiol. 2008 Apr;119(4):892-6. doi: 10.1016/j.clinph.2007.12.015. Epub 2008 Mar 4. PMID 18289932
- [Background] Dimitrijevic MM, Dimitrijevic MR, Illis LS, Nakajima K, Sharkey PC, Sherwood AM. Spinal cord stimulation for the control of spasticity in patients with chronic spinal cord injury: I. Clinical observations. Cent Nerv Syst Trauma. 1986 Spring;3(2):129-44. doi: 10.1089/cns.1986.3.129. PMID 3490312
- [Background] Dimitrijevic MR, Illis LS, Nakajima K, Sharkey PC, Sherwood AM. Spinal cord stimulation for the control of spasticity in patients with chronic spinal cord injury: II. Neurophysiologic observations. Cent Nerv Syst Trauma. 1986 Spring;3(2):145-52. doi: 10.1089/cns.1986.3.145. PMID 3490313
- [Background] Dobkin B, Apple D, Barbeau H, Basso M, Behrman A, Deforge D, Ditunno J, Dudley G, Elashoff R, Fugate L, Harkema S, Saulino M, Scott M; Spinal Cord Injury Locomotor Trial Group. Weight-supported treadmill vs over-ground training for walking after acute incomplete SCI. Neurology. 2006 Feb 28;66(4):484-93. doi: 10.1212/01.wnl.0000202600.72018.39. PMID 16505299
- [Background] Dy CJ, Gerasimenko YP, Edgerton VR, Dyhre-Poulsen P, Courtine G, Harkema SJ. Phase-dependent modulation of percutaneously elicited multisegmental muscle responses after spinal cord injury. J Neurophysiol. 2010 May;103(5):2808-20. doi: 10.1152/jn.00316.2009. PMID 20357075
- [Background] Einhorn J, Li A, Hazan R, Knikou M. Cervicothoracic multisegmental transpinal evoked potentials in humans. PLoS One. 2013 Oct 7;8(10):e76940. doi: 10.1371/journal.pone.0076940. eCollection 2013. PMID 24282479
- [Background] Field-Fote EC, Roach KE. Influence of a locomotor training approach on walking speed and distance in people with chronic spinal cord injury: a randomized clinical trial. Phys Ther. 2011 Jan;91(1):48-60. doi: 10.2522/ptj.20090359. Epub 2010 Nov 4. PMID 21051593
- [Background] Gad P, Choe J, Shah P, Garcia-Alias G, Rath M, Gerasimenko Y, Zhong H, Roy RR, Edgerton VR. Sub-threshold spinal cord stimulation facilitates spontaneous motor activity in spinal rats. J Neuroeng Rehabil. 2013 Oct 24;10:108. doi: 10.1186/1743-0003-10-108. PMID 24156340
- [Background] Hajela N, Mummidisetty CK, Smith AC, Knikou M. Corticospinal reorganization after locomotor training in a person with motor incomplete paraplegia. Biomed Res Int. 2013;2013:516427. doi: 10.1155/2013/516427. Epub 2012 Dec 26. PMID 23484130
- [Background] Hofstoetter US, Knikou M, Guertin PA, Minassian K. Probing the Human Spinal Locomotor Circuits by Phasic Step-Induced Feedback and by Tonic Electrical and Pharmacological Neuromodulation. Curr Pharm Des. 2017;23(12):1805-1820. doi: 10.2174/1381612822666161214144655. PMID 27981912
- [Background] Hofstoetter US, Krenn M, Danner SM, Hofer C, Kern H, McKay WB, Mayr W, Minassian K. Augmentation of Voluntary Locomotor Activity by Transcutaneous Spinal Cord Stimulation in Motor-Incomplete Spinal Cord-Injured Individuals. Artif Organs. 2015 Oct;39(10):E176-86. doi: 10.1111/aor.12615. Epub 2015 Oct 6. PMID 26450344
- [Background] Hofstoetter US, McKay WB, Tansey KE, Mayr W, Kern H, Minassian K. Modification of spasticity by transcutaneous spinal cord stimulation in individuals with incomplete spinal cord injury. J Spinal Cord Med. 2014 Mar;37(2):202-11. doi: 10.1179/2045772313Y.0000000149. Epub 2013 Nov 26. PMID 24090290
- [Background] Hofstoetter US, Minassian K, Hofer C, Mayr W, Rattay F, Dimitrijevic MR. Modification of reflex responses to lumbar posterior root stimulation by motor tasks in healthy subjects. Artif Organs. 2008 Aug;32(8):644-8. doi: 10.1111/j.1525-1594.2008.00616.x. PMID 18782137
- [Background] Hunanyan AS, Petrosyan HA, Alessi V, Arvanian VL. Repetitive spinal electromagnetic stimulation opens a window of synaptic plasticity in damaged spinal cord: role of NMDA receptors. J Neurophysiol. 2012 Jun;107(11):3027-39. doi: 10.1152/jn.00015.2012. Epub 2012 Mar 7. PMID 22402659
- [Background] James ND, Bartus K, Grist J, Bennett DL, McMahon SB, Bradbury EJ. Conduction failure following spinal cord injury: functional and anatomical changes from acute to chronic stages. J Neurosci. 2011 Dec 14;31(50):18543-55. doi: 10.1523/JNEUROSCI.4306-11.2011. PMID 22171053
- [Background] Knikou M. The H-reflex as a probe: pathways and pitfalls. J Neurosci Methods. 2008 Jun 15;171(1):1-12. doi: 10.1016/j.jneumeth.2008.02.012. Epub 2008 Mar 4. PMID 18394711
- [Background] Knikou M. Neural control of locomotion and training-induced plasticity after spinal and cerebral lesions. Clin Neurophysiol. 2010 Oct;121(10):1655-68. doi: 10.1016/j.clinph.2010.01.039. Epub 2010 Apr 27. PMID 20427232
- [Background] Knikou M. Plasticity of corticospinal neural control after locomotor training in human spinal cord injury. Neural Plast. 2012;2012:254948. doi: 10.1155/2012/254948. Epub 2012 Jun 4. PMID 22701805
- [Background] Knikou M. Neurophysiological characterization of transpinal evoked potentials in human leg muscles. Bioelectromagnetics. 2013 Dec;34(8):630-40. doi: 10.1002/bem.21808. Epub 2013 Sep 20. PMID 24115026
- [Background] Knikou M. Neurophysiological characteristics of human leg muscle action potentials evoked by transcutaneous magnetic stimulation of the spine. Bioelectromagnetics. 2013 Apr;34(3):200-10. doi: 10.1002/bem.21768. Epub 2012 Nov 28. PMID 23192827
- [Background] Knikou M. Functional reorganization of soleus H-reflex modulation during stepping after robotic-assisted step training in people with complete and incomplete spinal cord injury. Exp Brain Res. 2013 Jul;228(3):279-96. doi: 10.1007/s00221-013-3560-y. Epub 2013 May 25. PMID 23708757
- [Background] Knikou M. Transpinal and transcortical stimulation alter corticospinal excitability and increase spinal output. PLoS One. 2014 Jul 9;9(7):e102313. doi: 10.1371/journal.pone.0102313. eCollection 2014. PMID 25007330
- [Background] Knikou M, Angeli CA, Ferreira CK, Harkema SJ. Soleus H-reflex modulation during body weight support treadmill walking in spinal cord intact and injured subjects. Exp Brain Res. 2009 Mar;193(3):397-407. doi: 10.1007/s00221-008-1636-x. Epub 2008 Nov 15. PMID 19011843
- [Background] Knikou M, Angeli CA, Ferreira CK, Harkema SJ. Flexion reflex modulation during stepping in human spinal cord injury. Exp Brain Res. 2009 Jul;196(3):341-51. doi: 10.1007/s00221-009-1854-x. Epub 2009 May 26. PMID 19468720
- [Background] Knikou M, Conway BA. Effects of electrically induced muscle contraction on flexion reflex in human spinal cord injury. Spinal Cord. 2005 Nov;43(11):640-8. doi: 10.1038/sj.sc.3101772. PMID 15968304
- [Background] Knikou M, Dixon L, Santora D, Ibrahim MM. Transspinal constant-current long-lasting stimulation: a new method to induce cortical and corticospinal plasticity. J Neurophysiol. 2015 Sep;114(3):1486-99. doi: 10.1152/jn.00449.2015. Epub 2015 Jun 24. PMID 26108955
- [Background] Knikou M, Smith AC, Mummidisetty CK. Locomotor training improves reciprocal and nonreciprocal inhibitory control of soleus motoneurons in human spinal cord injury. J Neurophysiol. 2015 Apr 1;113(7):2447-60. doi: 10.1152/jn.00872.2014. Epub 2015 Jan 21. PMID 25609110
- [Background] Knikou M, Hajela N, Mummidisetty CK, Xiao M, Smith AC. Soleus H-reflex phase-dependent modulation is preserved during stepping within a robotic exoskeleton. Clin Neurophysiol. 2011 Jul;122(7):1396-404. doi: 10.1016/j.clinph.2010.12.044. Epub 2011 Jan 14. PMID 21237704
- [Background] Knikou M, Hajela N, Mummidisetty CK. Corticospinal excitability during walking in humans with absent and partial body weight support. Clin Neurophysiol. 2013 Dec;124(12):2431-8. doi: 10.1016/j.clinph.2013.06.004. Epub 2013 Jun 28. PMID 23810634
- [Background] Knikou M, Mummidisetty CK. Locomotor training improves premotoneuronal control after chronic spinal cord injury. J Neurophysiol. 2014 Jun 1;111(11):2264-75. doi: 10.1152/jn.00871.2013. Epub 2014 Mar 5. PMID 24598526
- [Background] Maertens de Noordhout A, Rothwell JC, Thompson PD, Day BL, Marsden CD. Percutaneous electrical stimulation of lumbosacral roots in man. J Neurol Neurosurg Psychiatry. 1988 Feb;51(2):174-81. doi: 10.1136/jnnp.51.2.174. PMID 2831302
- [Background] Maiman DJ, Mykleburst JB, Barolat-Romana G. Spinal cord stimulation for amelioration of spasticity: experimental results. Neurosurgery. 1987 Sep;21(3):331-3. doi: 10.1227/00006123-198709000-00008. PMID 3499582
- [Background] Minassian K, Hofstoetter US. Spinal Cord Stimulation and Augmentative Control Strategies for Leg Movement after Spinal Paralysis in Humans. CNS Neurosci Ther. 2016 Apr;22(4):262-70. doi: 10.1111/cns.12530. Epub 2016 Feb 18. PMID 26890324
- [Background] Minassian K, Hofstoetter US, Danner SM, Mayr W, Bruce JA, McKay WB, Tansey KE. Spinal Rhythm Generation by Step-Induced Feedback and Transcutaneous Posterior Root Stimulation in Complete Spinal Cord-Injured Individuals. Neurorehabil Neural Repair. 2016 Mar;30(3):233-43. doi: 10.1177/1545968315591706. Epub 2015 Jun 18. PMID 26089308
- [Background] Murray LM, Knikou M. Remodeling Brain Activity by Repetitive Cervicothoracic Transspinal Stimulation after Human Spinal Cord Injury. Front Neurol. 2017 Feb 20;8:50. doi: 10.3389/fneur.2017.00050. eCollection 2017. PMID 28265259
- [Background] Smith AC, Knikou M. A Review on Locomotor Training after Spinal Cord Injury: Reorganization of Spinal Neuronal Circuits and Recovery of Motor Function. Neural Plast. 2016;2016:1216258. doi: 10.1155/2016/1216258. Epub 2016 May 11. PMID 27293901
- [Background] Smith AC, Mummidisetty CK, Rymer WZ, Knikou M. Locomotor training alters the behavior of flexor reflexes during walking in human spinal cord injury. J Neurophysiol. 2014 Nov 1;112(9):2164-75. doi: 10.1152/jn.00308.2014. Epub 2014 Aug 13. PMID 25122715
- [Background] Smith AC, Rymer WZ, Knikou M. Locomotor training modifies soleus monosynaptic motoneuron responses in human spinal cord injury. Exp Brain Res. 2015 Jan;233(1):89-103. doi: 10.1007/s00221-014-4094-7. Epub 2014 Sep 10. PMID 25205562
- [Background] Thomas SL, Gorassini MA. Increases in corticospinal tract function by treadmill training after incomplete spinal cord injury. J Neurophysiol. 2005 Oct;94(4):2844-55. doi: 10.1152/jn.00532.2005. Epub 2005 Jul 6. PMID 16000519
- [Background] Wirz M, Zemon DH, Rupp R, Scheel A, Colombo G, Dietz V, Hornby TG. Effectiveness of automated locomotor training in patients with chronic incomplete spinal cord injury: a multicenter trial. Arch Phys Med Rehabil. 2005 Apr;86(4):672-80. doi: 10.1016/j.apmr.2004.08.004. PMID 15827916